CLINICAL TRIAL: NCT01732250
Title: Multicenter Open-label RCT to Compare Colistin Alone vs. Colistin Plus Meropenem
Brief Title: Multicenter Open-label Randomized Controlled Trial (RCT) to Compare Colistin Alone Versus Colistin Plus Meropenem
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mical Paul (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor-Investigator, Mical Paul, MD, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0276-12-RMC
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Gram-Negative Bacterial Infections
Keywords: Gram-Negative Bacterial Infections; Resistant Bacteria; Drug Resistance, Bacterial; Colistin
MeSH Terms: conditions — Gram-Negative Bacterial Infections | interventions — Colistin; colistinmethanesulfonic acid; Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colistin and Meropenem (Experimental): IV meropenem, 2 gram q8h, adjusted for renal function IV Colistin with loading dose of 9 mil IU units, Maintenance dose 4.5 mil IU q12h, adjusted for renal function
  Interventions: Drug: Colistin; Drug: Meropenem
- Colistin (Active Comparator): IV Colistin with loading dose of 9 mil IU units, Maintenance dose 4.5 mil IU q12h, adjusted for renal function
  Interventions: Drug: Colistin

INTERVENTIONS:
Drug: Colistin — IV Colistin with loading dose of 9 mil IU units, Maintenance dose 4.5 mil IU q12h, adjusted for renal function, for 10 days.
  Other Names: Colistimethate Sodium; Coliracin
Drug: Meropenem — IV meropenem, 2 gram q8h, adjusted for renal function, for up to 10 days.
  Other Names: Meronem
  Arms: Colistin and Meropenem

SUMMARY:
The purpose of this study is to determine whether the addition of meropenem to colistin is better than colistin alone in the treatment of clinically significant infections caused by multi-drug resistant bacteria

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients
* Clinically significant, microbiological-documented infection caused by carbapenem-resistant and colistin-susceptible Gram-negative bacteria and identified according to CDC criteria- blood stream infections, hospital acquired pneumonia, ventilator associated pneumonia, and urinary tract infections
* Patient recruitment will occur only after microbiological documentation and susceptibility testing. Patients will be included within 96 hours of the time the index culture was taken (typically within 48 hours of isolate identification), regardless of the antibiotic treatment administered during this time period.

Exclusion Criteria:

* Previous inclusion in the trial. Patients will be included in the RCT only once for the first identified episode of infection
* Pregnant women
* Epilepsy or prior seizures
* Known allergy to colistin or a carbapenem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Clinical success | 14 days
  defined as a composite of all of the following, all measured at 14 days:
  * Patient alive
  * Systolic blood pressure >90 mmHg without need for vasopressor support
  * Stable or improved SOFA score, define as:
    * for baseline SOFA ≥ 3: a decrease of at least 30%;
    * for baseline SOFA <3: stable or decreased SOFA score
  * For patients with HAP/ VAP, PaO2/FiO2 ratio stable or improved
  * For patients with bacteremia, no growth of the initial isolate in blood cultures taken on day 14 if patient still febrile

SECONDARY OUTCOMES:
Secondary outcomes and adverse events | 14 and 28 days
  14 and 28-day all-cause mortality.
  If patients are discharged or death occurs before end of follow-up (day 28), we will end data collection at that date. We will attempt to determine survival status at day 28 for all patients (central registry in Israel; re-admissions, rehabilitation centers, hospital transfers in Greece and Italy).
Clinical success with modification | 14 days
  Clinical success, but with modification to the antibiotic treatment not permitted by protocol
Time to defervescence | 28 days
  defined as time to reach a temperature of <38°C with no recurrence for 3 days
Time to weaning | 28 days
  Time to weaning from mechanical ventilation in VAP for patients weaned alive
Time to hospital discharge | 28 days
  Time to hospital discharge for patient discharged alive
Microbiological failure | 28 days
  Microbiological failure, defined as isolation of the initial isolate (phenotypically identical) in a clinical sample (blood or other) 7 days or more after start of treatment or its identification in respiratory samples.
  * For all patients with VAP/ HAP sputum or tracheal aspirates will be obtained on day 7, regardless of clinical response
  * For all patients with UTI, a repeat urine culture will be obtained on day 7, regardless of clinical response
  * For patients with bacteremia, blood cultures will be repeated on day 7 and 14, only if the patient is febrile at that time
Superinfections | 28 days
  Defined as a new clinically or microbiologically-documented infections by CDC criteria within 28 days
New resistant infection | 28 days
  Colonization or infection by newly-acquired (other species than the initial infection) carbapenem-resistant or colistin-resistant Gram-negative bacteria. Colonization will be assessed by rectal surveillance
CDAD | 28 days
  Clostridium-difficile-associated diarrhea, defined by diarrhea with a positive C. difficile toxin test

CONTACTS AND LOCATIONS:
Overall Officials: Johan Mouton, MD PhD, Study Chair — Radboud University Medical Center; Mical Paul, MD, Principal Investigator — Rambam Health Care Centre
Locations (7):
- Greece (2):
  - Atikkon Hospital, Athens
  - Laikon Hosptial, Athens
- Israel (3):
  - Rambam Health Care Center, Haifa
  - Rabin Medical Center, Petach-Tikvah
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Monaldi Hospital, University of Naples S.U.N., Naples
  - Agostino Gemelli Hospital, Rome

REFERENCES:
- [Derived] Nutman A, Temkin E, Lellouche J, Amar Ben Dalak M, Kaplan E, Lurie-Weinberger M, Dishon Benattar Y, Neuberger A, Stern A, Daitch V, Eliakim-Raz N, Durante-Mangoni E, Bernardo M, Iossa D, Daikos G, Skiada A, Pavleas I, Friberg L, Theuretzbacher U, Leibovici L, Paul M, Carmeli Y; AIDA Study Group. Carbapenem-resistant Enterobacterales (CRE) acquisition and molecular characterization following colistin monotherapy and colistin-meropenem combination therapy: findings from the AIDA randomized trial. Antimicrob Resist Infect Control. 2025 Nov 5;14(1):133. doi: 10.1186/s13756-025-01651-1. PMID 41194117
- [Derived] Daitch V, Paul M, Daikos GL, Durante-Mangoni E, Yahav D, Carmeli Y, Benattar YD, Skiada A, Andini R, Eliakim-Raz N, Nutman A, Zusman O, Antoniadou A, Cavezza G, Adler A, Dickstein Y, Pavleas I, Zampino R, Bitterman R, Zayyad H, Koppel F, Zak-Doron Y, Levi I, Babich T, Turjeman A, Ben-Zvi H, Friberg LE, Mouton JW, Theuretzbacher U, Leibovici L. Excluded versus included patients in a randomized controlled trial of infections caused by carbapenem-resistant Gram-negative bacteria: relevance to external validity. BMC Infect Dis. 2021 Mar 31;21(1):309. doi: 10.1186/s12879-021-05995-y. PMID 33789574
- [Derived] Dickstein Y, Lellouche J, Ben Dalak Amar M, Schwartz D, Nutman A, Daitch V, Yahav D, Leibovici L, Skiada A, Antoniadou A, Daikos GL, Andini R, Zampino R, Durante-Mangoni E, Mouton JW, Friberg LE, Dishon Benattar Y, Bitterman R, Neuberger A, Carmeli Y, Paul M; AIDA Study Group. Treatment Outcomes of Colistin- and Carbapenem-resistant Acinetobacter baumannii Infections: An Exploratory Subgroup Analysis of a Randomized Clinical Trial. Clin Infect Dis. 2019 Aug 16;69(5):769-776. doi: 10.1093/cid/ciy988. PMID 30462182
- [Derived] Paul M, Daikos GL, Durante-Mangoni E, Yahav D, Carmeli Y, Benattar YD, Skiada A, Andini R, Eliakim-Raz N, Nutman A, Zusman O, Antoniadou A, Pafundi PC, Adler A, Dickstein Y, Pavleas I, Zampino R, Daitch V, Bitterman R, Zayyad H, Koppel F, Levi I, Babich T, Friberg LE, Mouton JW, Theuretzbacher U, Leibovici L. Colistin alone versus colistin plus meropenem for treatment of severe infections caused by carbapenem-resistant Gram-negative bacteria: an open-label, randomised controlled trial. Lancet Infect Dis. 2018 Apr;18(4):391-400. doi: 10.1016/S1473-3099(18)30099-9. Epub 2018 Feb 16. PMID 29456043
- [Derived] Dickstein Y, Leibovici L, Yahav D, Eliakim-Raz N, Daikos GL, Skiada A, Antoniadou A, Carmeli Y, Nutman A, Levi I, Adler A, Durante-Mangoni E, Andini R, Cavezza G, Mouton JW, Wijma RA, Theuretzbacher U, Friberg LE, Kristoffersson AN, Zusman O, Koppel F, Dishon Benattar Y, Altunin S, Paul M; AIDA consortium. Multicentre open-label randomised controlled trial to compare colistin alone with colistin plus meropenem for the treatment of severe infections caused by carbapenem-resistant Gram-negative infections (AIDA): a study protocol. BMJ Open. 2016 Apr 20;6(4):e009956. doi: 10.1136/bmjopen-2015-009956. PMID 27098822